CLINICAL TRIAL: NCT03966495
Title: Sustainability of a Research Program in Risk Management: Routine Implementation, Appropriation, Effectiveness, Development of the Safety Culture
Brief Title: Sustainability of a Research Program in Risk Management (PeRENNITe)
Acronym: SUSTAIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0043
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: RM Program
MeSH Terms: interventions — Risk Management

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PRisM program: Pluriprofessional primary care offices with the PRiSM RM program:
  * Nine of the pluriprofessional primary care offices which implemented the RM program tested in the PRiSM study (2015-2017). The program consisted in: 1) Training on RM in the context of primary care; 2) The appointment of a RM referent in the office; 3) The conduct of six incident review meetings.
  * All participating offices had to declare adverse events that occurred during the time frame of the PRiSM study.
  * All participating offices had to fill in the safety climate survey MOSPS at the beginning and at the end of the PRiSM study.
  Interventions: Other: Sustainability of a research program in risk management
- Control: Pluriprofessional primary care offices without the PRiSM RM program:
  * Nine of the offices pluriprofessional primary care offices which didn't implement the RM program tested in the PRiSM study (2015-2017). They belonged to the PRisM study control group.
  * All participating offices had to declare adverse events that occurred during the time frame of the PRiSM study.
  * All participating offices had to fill in the safety climate survey MOSPS at the beginning and at the end of the PRiSM study.
  Interventions: Other: Sustainability of a research program in risk management

INTERVENTIONS:
Other: Sustainability of a research program in risk management — No intervention will be implemented in the present study.
  The investigators will evaluate of the sustainability of a research program in risk management in pluriprofessional primary care offices:
  * Qualitatively assessed safety culture and Sustainability of the PRisM RM program in the offices by interviews of professional belonging to the offices.
  * Quantitatively assessed safety climate in the offices measured by the Medical Office Survey on Patient Safety Culture (MOSPS) Questionnaire (fill in by the professionals of the offices)

SUMMARY:
Sustainability can be defined by several dimensions: the pursuit of program elements, the maintenance of its effectiveness, its integration into work processes, the adaptation of the program to the local context, its integration into the organizational culture, the dissemination of the program to other centres. Studies show that the continuation of the entire intervention is rare once the research stops.

The PRisM study (Pluriprofessionality and Risk Management through a Multifaceted Program in Primary Care) was a primary care risk management (RM) research project. Its purpose was to develop a safety culture within the participating multi-professional primary care structures. From 2015 to 2017, multi-professional primary care offices participated in the study, half of which implemented a RM program consisting of: 1) Training on RM in the context of primary care; 2) The appointment of a RM referent; 3) The conduct of six meetings of systematic analysis of incidents.

The PRisM study represents a favorable ground for the development of a methodology for evaluating the sustainability of a RM program in primary care.

ELIGIBILITY:
Inclusion Criteria:

* Volontary pluriprofessional primary care offices
* Having participated in the PRiSM study

Exclusion Criteria:

* office that waived participation in the PRisM study course
* office with a participation rate in the first PRisM safety climate survey < 30%.
* office of the PRisM study intervention group that did not implement the program as planned

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pluriprofessional primary care offices in France (called "centre, pôle et maison de santé pluridisciplinaire")
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
patient safety culture | 24 months from the end of the PRiSM study in 2017 (2019)
  - Qualitatively assessed through the model developed for health by Reiman, which apprehends the safety culture through organizational dimensions, social processes and psychological dimensions
patient safety culture | 24 months from the end of the PRiSM study in 2017 (2019)
  - Quantitatively assessed through 13 safetyclimate dimensions measured by the Medical Office Survey on Patient Safety Culture (MOSPS) Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Pauline OCCELLI, MD, Study Director — Hospices Civils de Lyon
Locations (1):
- Pôle de Santé publique des HCL, Lyon, France